CLINICAL TRIAL: NCT05344560
Title: Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-Energy Visible Light Produced on Commercial Manufacturing Lines
Brief Title: Evaluation of Toric Soft Contact Lenses Containing a Chromophore to Block High-Energy Visible Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6484
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Visual Acuity
MeSH Terms: interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- test/control/control (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (test/control/control) sequence and will wear two different study lenses one at a time bilaterally over three wear periods.
  Interventions: Device: soft contact lens in senofilcon A (C3) with HEVL-blocking chromophore; Device: ACUVUE OASYS 1-Day for Astigmatism
- control/test/test (Experimental): Eligible subjects that are habitual contact lens wearers will be randomized into the (control/test/test) sequence and will wear two different study lenses one at a time bilaterally over three wear periods.
  Interventions: Device: soft contact lens in senofilcon A (C3) with HEVL-blocking chromophore; Device: ACUVUE OASYS 1-Day for Astigmatism

INTERVENTIONS:
Device: soft contact lens in senofilcon A (C3) with HEVL-blocking chromophore — TEST Lens
Device: ACUVUE OASYS 1-Day for Astigmatism — CONTROL Lens

SUMMARY:
This will be a 4-visit, randomized, controlled, single-masked, bilateral wear, dispensing, 2-treament, 2-sequence, 3-period crossover study to evalulate overall vision and comfort..

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy of all the following criteria to be enrolled in the study.

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 years of age (inclusive) at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily or daily disposable wear modality (i.e. not extended wear modality). Habitual wearer is defined as a minimum of 6 hours per day, for a minimum of 2 days per week during the past four weeks.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study:

   1. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps
   2. Cylinder powers (DC) -0.75 and -1.25
   3. Axes (degrees) 170, 180, 10, 80, 90, 100
7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have an ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (10):
- United States (10):
  - Dr. James Weber & Associates, PA - City Square Blvd, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Southwest Orlando Eye Care, Orlando, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - ProCare Vision Centers, Granville, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island
  - Optometry Group, LLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 subjects were enrolled in this study. Of those enrolled, all 126 subjects were dispensed at least one study lens. Of those dispensed, 119 subjects completed the study while 7 subjects were discontinued.
Groups:
- Test\Control\Control: Subjects in this sequence were randomized to receive the Test [senofilcon A (C3) HEV chromophore] lens during the first period and the Control [senofilcon A (C3)] lens during the second and third periods .
- Control\Test\Test: Subjects in this sequence were randomized to receive the Control [senofilcon A (C3)] lens during the first period and the Test [senofilcon A (C3) HEV chromophore] lens during the second and third periods.
Period: Period 1
Arm/Group | Test\Control\Control | Control\Test\Test
Started | 63 | 63
Completed | 62 | 62
Not Completed | 1 | 1
Not completed — Subject out of visit window | 1 | 1
Period: Period 2
Arm/Group | Test\Control\Control | Control\Test\Test
Started | 62 | 62
Completed | 59 | 61
Not Completed | 3 | 1
Not completed — Covid-19 Related | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Subject out of visit window | 1 | 1
Period: Period 3
Arm/Group | Test\Control\Control | Control\Test\Test
Started | 59 | 61
Completed | 58 | 61
Not Completed | 1 | 0
Not completed — Subject out of visit window | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 41
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3
  Black or African American | 11
  White | 111
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 126

OUTCOME MEASURES:

1. Primary Outcome: CLUE Comfort Score
Description: Subjective comfort was assessed using Contact Lens User Experience (CLUE) questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (Comfort, Vision, Handling, and Packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution where scores range from 0 to 120 with a population average score of 60 (SD 20). Higher CLUE scores indicate a more favorable/positive response. The average CLUE comfort score was report for each lens type.
Time Frame: 1-Week Follow-up
Population: All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Test [Senofilcon A (C3) HEV Chromophore]: Subjects that wore the Test [senofilcon A (C3) HEV chromophore] lens during any of the three study periods.
- Control [Senofilcon A (C3)]: Subjects that wore the Control [senofilcon A (C3)] lens during any of the three study periods.
Arm/Group | Test [Senofilcon A (C3) HEV Chromophore] | Control [Senofilcon A (C3)]
Number analyzed (Participants) | 119 | 119
Units on a scale | 63.50 (19.581) | 65.28 (20.915)
Statistical Analysis 1: Comparison: Test [Senofilcon A (C3) HEV Chromophore] vs Control [Senofilcon A (C3)]; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-6.92 to 1.07], Standard Error of Mean 2.018 — Mean difference was calculated as Test [senofilcon A (C3) HEV chromophore] minus Control [senofilcon A (C3)]

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; Approximately 3-weeks per subject.
Groups:
- Test [Senofilcon A (C3) HEV Chromophore]: Subjects that wore the Test [senofilcon A (C3) HEV chromophore] lens during any point in the study.
- Control [Senofilcon A (C3)]: Subjects that wore the Control [senofilcon A (C3)] lens during any point in the study.
Arm/Group | Test [Senofilcon A (C3) HEV Chromophore] | Control [Senofilcon A (C3)]
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/125
Other Adverse Events (participants affected / at risk) | 0/125 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT05344560/Prot_SAP_000.pdf